CLINICAL TRIAL: NCT02124278
Title: A Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of PUL-042 Inhalation Solution in Healthy Subjects
Brief Title: Safety and Tolerability of Single Ascending Doses of PUL-042 Inhalation Solution in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pulmotect, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PUL-042-001
Record Dates: First submitted 2014-04-24; First posted 2014-04-28 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Healthy
Keywords: Single ascending dose; Safety and tolerability in healthy subjects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PUL-042 Inhalation Solution (Experimental): Fixed dose combination of Pam2CSK4 acetate (Pam2) and ODN M362 (ODN) administered as an inhalation solution. Single dose administration by nebulization. Starting dose will be 2.9 micrograms Pam2: 4.25 micrograms ODN. Up to 7 doubling doses may be tested.
  Interventions: Drug: PUL-042 Inhalation Solution
- Sterile water for injection (Placebo Comparator): Sterile water for injection administered by nebulization
  Interventions: Drug: PUL-042 Inhalation Solution

INTERVENTIONS:
Drug: PUL-042 Inhalation Solution

SUMMARY:
The purpose is to determine if single doses of PUL-042 inhalation solution are safe in healthy subjects.

DETAILED DESCRIPTION:
The study will assess the safety, tolerability, pharmacokinetics and pharmacodynamics of single ascending doses of PUL-042 inhalation solutions in healthy subjects.

Subjects will be enter a screening period of up to 14 days to determine eligibility. Subjects will be admitted to the Phase 1 unit the day prior to dosing and remain in the unit until 24 hours post-dose. Subjects will be seen in the clinic at 3 and 7 days post-dose

A modified 3+3 design will be used to determine the maximum tolerated dose (MTD) based on the occurrence of dose-limiting toxicities (DLTs) defined by Common Terminology Criteria for Adverse Events (CTCAE) v4. Additional specific DLTs will be defined as: 1) Hypoxia, defined as a non-artifactual drop in pulse oximetry to < 90% on room air, 2) A decrease in forced expiratory volume in one second (FEV1) of 12% or greater compared to the last observation prior to dosing, 3) Any evidence of bronchospasm or wheezing requiring medical intervention. Doses will be doubled until the maximum tolerated dose (MTD- defined as the largest dose with 0/6 or 1/6 DLTs) is reached.

ELIGIBILITY:
Inclusion Criteria:

* Males or females of non-childbearing potential
* Body mass index between 18 and 30 kg/m2
* Normal spirometry
* Normal diffusing capacity of lung for carbon monoxide
* Normal pulse oximetry
* Males willing to practice contraception or have a female partner using contraception

Exclusion Criteria:

* Febrile
* Abnormal chest x-ray
* History of tobacco products within the last year and total exposure of > 5 pack/years
* Clinically significant laboratory findings
* History of chronic pulmonary disease
* History of atopic reactions
* Mediastinal lymphadenopathy
* Oral corticosteroid therapy within 4 weeks prior to randomization
* Alcohol, caffeine or strenuous exercise within 72 hours prior to dosing
* Grapefruit within 7 days prior to dosing
* Administration of concomitant medications within 14 days prior to dosing
* Exposure to any investigational agent with 30 days
* Significant concurrent illness
* Know positive for HIV, hepatitis B or hepatitis C
* Inability to tolerate a nebulization test with sterile water for injection
* Positive test for drugs of abuse

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2014-02; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicities (DLTs) | Dosing to one week post-dose

CONTACTS AND LOCATIONS:
Locations (1):
- ICON Development Solutions, San Antonio, Texas, United States